CLINICAL TRIAL: NCT00401804
Title: Bortezomib-Doxorubicin-Dexamethasone as Treatment for Patients With Multiple Myeloma Presenting With Acute Renal Failure
Brief Title: Bortezomib-Dexamethasone-Doxorubicin-Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Austrian Forum Against Cancer (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Eudract Number: 2005-003001-85
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2010-07

CONDITIONS: Multiple Myeloma; Renal Insuficiency
Keywords: Multiple Myeloma; renal impairment; Velcade
MeSH Terms: conditions — Multiple Myeloma; Renal Insufficiency | interventions — Dexamethasone; Bortezomib; Doxorubicin

INTERVENTIONS:
Drug: Dexamethasone, Bortezomib, Doxorubicin

SUMMARY:
The primary objective of the study is to evaluate the activity of BDD in subjects with acute renal failure as measured by· reversal of acute renal failureSecondary objectives· tumor response (complete and partial response)· To evaluate the safety of Bortezomib- Doxorubicin-Dexamethasone in this patient population· to evaluate the activity of Bortezomib- Doxorubicin -Dexamethasone on progression free survival · to evaluate the activity of Bortezomib- Doxorubicin -Dexamethasone on overall survival

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple myeloma ·
* Acute multiple myeloma related renal failure (Diagnosis established by clinical and laboratory findings including renal biopsy - if indicated)a) Newly diagnosed patients:Decrease of GFR to < 50ml/minb) Previously treated patients with GFR of ≥ 60ml/min within last 4 weeks: decrease in GFR > 25% and to < 60ml / min,concomitantly with either increase in paraproteins (>25%) and/or decrease in hemoglobin ≥ 2 g/dl (within 4 weeks) and/or increase in bone marrow plasma infiltration and/or increase in number of bone lesions and/or hypercalcaemia (Ca > 11.5 mg/dl or 2.8 mmol/l) as signs of disease progression·
* Age > 20 years·
* ECOG performance status of ≤ 3.·
* Platelet count > 50.000/µl·
* WBC > 2000/µl·
* Total bilirubin < 1.5 x upper limit of normal,
* AST, ALT < 2.5 x upper limit of normal·
* International Normalized Ratio (INR) < 1.5; APTT < 1.5 x upper limit of normal·
* Fertile women and men of childbearing potential (<2 years after last menstruation in women) must use effective means of contraception (oral contraceptives, intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly or surgically sterile)· Negative serum or urine β-HCG pregnancy test at screening for subjects of child-bearing potential·
* Patient's written informed consent

Exclusion Criteria:

* History of malignancy other than squamous cell carcinoma, basal cell carcinoma of the skin or carcinoma in situ of the cervix within the last 5 years.·
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study.·
* Evidence of CNS involvement or spinal cord compression.·
* Neuropathy Grade ≥ 2·
* A history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant and adversely affecting compliance to study drug.·
* NYHA Status > 2, i.e. clinically significant cardiac disease, (congestive heart failure, symptomatic coronary artery disease, cardiac arrhythmias, and arterial hypertension not well controlled with medication) or myocardial infarction within the last 6 months ·
* Evidence of bleeding diathesis or coagulopathy·
* Serious, non-healing wound or ulcer·
* Evidence of any severe active acute or chronic infection.·
* Evidence of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or patient at high risk from treatment complications·
* Patient is known to be HIV-positive, Hbs-antigen positive or HCV-RNA-positive·
* Pregnant women or nursing mothers·
* Have received bortezomib within 4 weeks before enrollment·
* Half body irradiation < 28 days before enrollment·
* Has known or suspected hypersensitivity or intolerance to boron, mannitol, or heparin, if an indwelling catheter is used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2006-02; Primary Completion 2008-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
OS

SECONDARY OUTCOMES:
OR

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Ludwig, MD, Univ.Prof., Principal Investigator — Austrian Forum agianst Cancer; Wilhelminenspital Vienna, 1st. Med. Department - center for Oncology and Hematology
Locations (9):
- Austria (8):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Klinischen Abteilung für Hämatologie, Medizinische Universitätsklinik Graz, Graz
  - Landeskrankenhaus Leoben, Leoben
  - Dep. of Internal Medicine I, Oncology, SALK - Gemeinnützige Salzburger Landeskliniken, Salzburg
  - Medical University of Vienna, Dep. of Internal Medicine I, Vienna
  - Universitätsklinik für Innere Medizin I, Vienna
  - Wilhelminenspital Vienna, 1st Med. Department - center for Oncology and Hematology, Vienna
  - Klinikum Kreuzschwestern Wels GmbH, Wels
- FN Brno Interni Hematoonkolog. klinika, Brno, Czechia

REFERENCES:
- [Derived] Ludwig H, Adam Z, Hajek R, Greil R, Tothova E, Keil F, Autzinger EM, Thaler J, Gisslinger H, Lang A, Egyed M, Womastek I, Zojer N. Light chain-induced acute renal failure can be reversed by bortezomib-doxorubicin-dexamethasone in multiple myeloma: results of a phase II study. J Clin Oncol. 2010 Oct 20;28(30):4635-41. doi: 10.1200/JCO.2010.28.1238. Epub 2010 Sep 7. PMID 20823423